CLINICAL TRIAL: NCT05204719
Title: Prophylactic Delivery Room Continuous Positive Airway Pressure to Optimize Outcomes in Spontaneously Breathing Late Preterm Neonates Born by Cesarean Section: A Pilot Clinical Trial
Brief Title: Prophylactic DR-CPAP on Late Preterm Infants Born by C-section: an RCT
Acronym: PLANT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other); Columbia University (Other); St. Louis University (Other); University of Alberta (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13965
Record Dates: First submitted 2021-11-23; First posted 2022-01-24 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Premature Birth
Keywords: Neonatal Resuscitation; Clinical Trial; Late Preterm Infants; Lung Aeration; Respiratory Transition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Delivery Room Continuous Positive Airway Pressure (Experimental): If the infant is spontaneously breathing and allocated to the experimental arm, s/he will receive 20 min of 5 cm H2O of prophylactic continuous airway pressure using either a face mask or the appropriate size of nasal prong.
  Interventions: Procedure: Prophylactic Delivery Room Continuous Positive Airway Pressure
- No Prophylactic Delivery Room Continuous Positive Airway Pressure (No Intervention): Alternatively, spontaneously breathing infants assigned to control group will receive the standard of care with no prophylactic delivery room continuous positive airway pressure (CPAP).
  In both groups, CPAP can be used to help babies with persistent labored breathing or cyanosis after the initial steps as per the participating institution's neonatal resuscitation protocol. At any time, if the patient does not present spontaneous breathing, an escalation on the resuscitation measures will be performed and the study intervention will be terminated.

INTERVENTIONS:
Procedure: Prophylactic Delivery Room Continuous Positive Airway Pressure — Prophylactic Delivery Room Continuous Positive Airway Pressure (DR-CPAP) of 5-6 cm H20 will be provided for 20 minutes through the face mask or the appropriate size of nasal prong after the initial steps as per the participating institution's neonatal resuscitation protocol.
  Other Names: DR-CPAP
  Arms: Prophylactic Delivery Room Continuous Positive Airway Pressure

SUMMARY:
A Pragmatic Randomized Controlled Pilot Trial to Evaluate the Impact of Early Prophylactic Continuous Positive Airway Pressure with or without Supplemental Oxygen in Spontaneously Breathing Late Preterm Newborn Infants Born by Cesarean Delivery, Compared to No Early Prophylactic Continuous Positive Airway Pressure with or without Supplemental Oxygen, on the Need for Further Respiratory Support Leading to NICU Admissions.

DETAILED DESCRIPTION:
A prospective multicenter randomized controlled trial of prophylactic delivery room continuous positive airway pressure (DR-CPAP) versus no prophylactic DR-CPAP will be conducted. Neonates with an obstetrically determined gestational age (GA) from 34 0/7 to 36 6/7 weeks born by Cesarean section (C-section) will be included. Patients to be screened will be identified from the electronic medical record by study personnel or by phone call from admitting physicians or obstetrics (OB) staff. In addition, a research nurse will screen and identify eligible women who are admitted to the OB service daily including labor and delivery or antepartum unit.

Eligible women will be approached by a trained research nurse about voluntary participation. If the patient is eligible the study will be introduced by research nurses independent of the treating or admitting physicians, and they will be provided with an informed consent form. Interested participants will be consented either on the antepartum unit or the labor and delivery unit prior to C-section. A total of 120 neonates will be enrolled in the trial, 60 in each group. Since mothers will be randomized to their respective groups immediately prior to C-section, twins will be allocated to the same treatment. The study will include neonates of both sexes and from all racial and ethnic groups. After obtaining the informed consent the research personnel will complete the eligibility electronic form including the information needed for the stratification (in the central web based system, Research Electronic Data Capture (REDCap) housed in a secure server. The central REDCap system will provide the group allocation.

The neonatal resuscitation team will ensure the required facemask or nasal prongs and the T piece resuscitator are available before delivery. Once the baby is born, the cord will be clamped following local practice and its time will be recorded. Then the initial steps following neonatal resuscitation guidelines will be performed (warming, drying, stimulating, positioning and suctioning if needed). An immediate evaluation of the respiratory status will be performed. If the infant is spontaneously breathing and allocated to the intervention group, they will receive 20 min of 5 to 6 cm water of continuous airway pressure using either a face mask or the appropriate size of nasal prong. Alternatively, spontaneously breathing infants assigned to control group will receive the standard of care with no prophylactic DR-CPAP. In both groups, CPAP can be used to help babies with persistent labored breathing or cyanosis after the initial steps as per the participating institutional neonatal resuscitation protocol. At any time, if the patient does not present spontaneous breathing, an escalation on the resuscitation measures will be performed and the study intervention will be terminated. A disposable pulse oximeter sensor of the appropriate size will be applied to the right wrist or hand as soon as possible. Supplemental oxygen will be provided to achieve the target oxygen saturation following neonatal resuscitation guidelines. Following delivery room management, all care decisions, including NICU admission, will be at discretion of the clinical team.

Participant data will be collected from the electronic medical record and/or from the monitoring equipment used during resuscitation (e.g., body temperature monitor, CPAP settings, and oxygen saturation, etc.). Patient characteristics, delivery room variables, and neonatal outcomes will be recorded in a secure password protected REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* Inborn newborns delivered by Cesarean section, gestational age between 34 weeks and < 37 weeks.

Exclusion Criteria:

* Major congenital anomalies including pulmonary hypoplasia and lethal life-limiting conditions.

Ages: 1 Minute to 5 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | up to 30 days or hospital discharge
  Duration of respiratory support including supplemental oxygen
Adverse outcomes | first 24 hours after birth
  Proportion of air leaks and any other safety related adverse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Birju A Shah, MD, Principal Investigator — Univeristy of Oklahoma Health Sciences Center
Locations (5):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Saint Louis University, St Louis, Missouri
  - The University of Oklahoma Health Campus, Oklahoma City, Oklahoma
- University of Alberta, Edmonton, Alberta, Canada
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah BA, Fabres JG, Leone TA, Schmolzer GM, Szyld EG; International Liaison Committee on Resuscitation Neonatal Life Support Task Force. Continuous positive airway pressure for term and >/=34+0 weeks' gestation newborns at birth: A systematic review. Resusc Plus. 2022 Nov 8;12:100320. doi: 10.1016/j.resplu.2022.100320. eCollection 2022 Dec. PMID 36386766